CLINICAL TRIAL: NCT02606734
Title: DyeVert Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osprey Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-6463
Record Dates: First submitted 2015-10-28; First posted 2015-11-17 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Angiography
MeSH Terms: interventions — Coronary Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Other): All subjects enrolled in the trial will use the DyeVert System.
  Interventions: Device: Coronary Angiography

INTERVENTIONS:
Device: Coronary Angiography — The DyeVert System will be used during coronary angiographic procedures which include: diagnostic only, diagnostic + PCI or PCI only cases.

SUMMARY:
The purpose of this study is to evaluate the usability characteristics of DyeVert™ during normal clinical use and to understand the amount of contrast media (CM) diverted from the subject and saved over a total angiographic procedure.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is indicated for a coronary angiogram or percutaneous coronary procedure
2. The subject is ≥ 18 years of age
3. The subject (or subject's legal representative) is willing and able to provide appropriate informed consent.

Exclusion Criteria:

1. Subject is undergoing a STEMI procedure
2. The subject is female and currently pregnant
3. In the investigator's opinion, the subject is not considered to be a suitable candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Monash Health, Clayton, Victoria, Australia
- University Hospital of Schleswig-Holstein, Lübeck, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Enrollment on 10/26/2015, Last Enrollment on 11/19/2015
Pre-assignment Details: Subjects undergoing a coronary artery imaging (angiogram) for diagnostic or percutaneous coronary intervention (PCI) procedures are eligible to participate in this study. All data will be collected on the day of the procedure. There are no follow-up visits in this study.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Australia | 20
  Germany | 24

OUTCOME MEASURES:

1. Primary Outcome: Volume (Percentage) of Contrast Media (CM) Diverted (Saved) in a Total Procedure
Description: The subject is exited from the study once they are discharged.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: percent of contrast media saved
Arm/Group | Treatment Arm
Number analyzed (Participants) | 44
percent of contrast media saved | 47.4 (8.7)

ADVERSE EVENTS:
Time Frame: AE Reporting occurred through the subjects discharge from the index procedure.
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No